CLINICAL TRIAL: NCT02786420
Title: Imaging Innovations for Placental Assessment in Response to Environmental Pollution
Brief Title: Imaging Innovations for Placental Assessment in Response to Environmental Pollution (PARENTs)
Acronym: PARENTs
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sherin Devaskar, Distinguished Professor of Pediatrics, Mattel Executive Endowed Chair, Department of Pediatrics, Executive Director, UCLA Children's Discovery and Innovation Institute, University of California, Los Angeles
Other Study IDs: 15-001388
Record Dates: First submitted 2016-04-14; First posted 2016-06-01 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Placental Disease
Keywords: pregnancy; magnetic resonance imaging; environmental air pollutants
MeSH Terms: conditions — Placenta Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen samples of blood and urine will be kept for further study related to this project involving markers relevant to placental insufficiency that may be discovered in the future. A gross assessment of the placenta will be performed by weighing the disc with cord and membranes removed. Cord insertion, length, diameter, coiling, number of vessels, focal lesions, membrane color, thickness, translucency, attachment, disc dimensions, range of thickness, fetal surface vascular distribution, pigmentation and site of rupture will be recorded. Microscopic assessment of H&E stained sections will be performed to detect any inflammatory/infectious processes, villous development/maturity, decidual vasculopathy, infarct/fibrin deposition, or other processes that may be associated with placental insufficiency and fetal development.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Pregnant women

SUMMARY:
How environmental pollution contributes to poor pregnancy outcome is poorly understood. The first trimester of pregnancy is a particularly vulnerable time period for the developing fetus and a mother's exposure to air pollution may alter the way that the placenta is established and how it functions throughout the rest of pregnancy. This project aims to expand and develop new MRI technologies to assess real-time placental structure and function as pregnancy develops from the first to the third trimester so that early detection, prevention strategies, and early treatment of placental dysfunction as a result of pollution exposures may be developed.

DETAILED DESCRIPTION:
Many epidemiological studies have associated exposure to traffic-derived air pollution from motor vehicles, air toxins from industry and other environmental toxins by pregnant women with measures of poor birth outcomes including preeclampsia (PE), preterm birth (PTB) and intra-uterine growth restriction (IUGR). Preeclampsia, preterm labor and IUGR, collectively known as ischemic placental disease, are strongly correlated with infant morbidity and a host of adult diseases ranging from coronary artery disease to cancer. Although it is widely believed that the pathophysiological mechanisms leading to complications of ischemic placental disease and placental insufficiency have similar biological origins, starting as early as defective placental implantation, to date there are no predictive studies that prospectively examine placental structure and/or function. This may be related to existing technologies, routinely employed in clinical decision-making, such as ultrasonography and certain biomarkers, lacking precision in the first trimester, and adequate sensitivity and specificity in the second to third trimesters. Thus, assessment and prediction of normalcy versus aberrancy of placental function are lacking. Therefore, the overarching objective of this proposal is to develop and evaluate a suit of cutting-edge multi-parametric magnetic resonance imaging (mp-MRI) technologies (primary predictor), and translate these novel placental imaging modalities to assessing the impact of environmental pollution exposure on prediction of the composite of placental aberrancy/insufficiency and related outcomes (PE, PTB and IUGR) (primary outcome).

Our central hypothesis is that chronic exposure to high rates of environmental pollution, independent of socio-economic status (SES), increases the risk of placental insufficiency due to early gestational development of adverse placental structure/function as detected by mp-MRI technological advances.

To test this hypothesis, our interdisciplinary research team at UCLA will first develop non-contrast freebreathing placental mp-MRI, consisting of multi-delay pseudo-continuous arterial spin labeling (pCASL) perfusion and high-resolution multi-contrast structural MRI, which will provide reproducible measures of placental perfusion and tissue microstructure (AIM 1). The novel mp-MRI techniques will be compared to the uterine artery Doppler ultrasound through pregnancy and validated ultimately by the gold standard histological pathology and vascularity of the post-parturient placenta (AIM 2). Lastly, the investigators will perform in-depth analyses of recruited subjects for exposure to environmental pollution and correlate their rates of exposure to extensively collected pregnancy outcomes, towards building a predictive model (AIM 3). Our specific aims are:

AIM 1: Develop non-contrast free-breathing placental mp-MRI techniques that can non-invasively characterize the in vivo placental perfusion and microstructure through all trimesters.

A. Develop a free-breathing multi-delay pCASL sequence using background-suppressed localized-volume 3D GRASE imaging for quantitative measurement of placental perfusion within a 5-10 min scan (1.5x1.5x2 mm3 resolution).

B. Develop a free-breathing high-resolution golden-angle 3D stack-of-radial sequence with self-navigation and retrospective motion compensation using compressed sensing for mapping placental microstructure within a 5-10 min scan (1x1x1 mm3 isotropic resolution).

AIM 2: Evaluate placental mp-MRI by longitudinal comparison with uterine artery Doppler ultrasound through gestation as a predictive marker of placental insufficiency.

A. Conduct a 3-year prospective cohort study of pregnant women, performing newly developed mp-MRI (AIM1) in the 1st and 2nd trimesters in parallel to ultrasound measurement of uterine artery Doppler, to assess mp-MRI prediction capability versus ultrasound.

B. Collect detailed pregnancy outcome data of prospective cohort, including diagnosis, neonatal outcome, and placenta for pathological and histological analysis to ascertain risk factors for placental insufficiency as a response to environmental exposures (AIM 3).

AIM 3: Perform in-depth analyses in recruited subjects to determine associations of environmental pollution exposures and both placental mp-MRI measurements and concomitant pregnancy outcomes.

A. Perform in-depth analyses to measures of modeled environmental pollution exposure in our recruited subjects to assess associations with mp-MRI measures of placental structure and perfusion throughout gestation, taking into account multiple confounding factors such as maternal age at delivery, race/ethnicity, and SES.

B. Correlate mp-MRI measures of placental structure and perfusion throughout gestation with pregnancy outcomes, post-parturient assessment of placental weight, pathology, and neonatal outcomes. These studies will establish the impact of environmental pollution on placental structure and function, and related pregnancy outcomes, with obstetric and neonatal practices embracing surveillance tactics based on the residential location of pregnant women and their offspring. In addition, the proposed research will establish the potential for early recognition of placental insufficiency, thereby staging future strategies of preventive and interventional therapies targeting reversal before encountering detrimental consequences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Planning to delivery at a UCLA hospital
* Carrying a viable pregnancy
* Not carrying multiple gestation

Exclusion Criteria:

* Known fetal chromosomal or structural abnormalities
* Contraindications to having MRI evaluation
* Inability to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Currently pregnant women who meet following eligibility criteria below
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-10-03 (Actual)

PRIMARY OUTCOMES:
Ischemic Placental Disease and Environment | 11 Weeks Gestational Age - Delivery
  To use multi-parametric MRI technology to assess the impact of environment pollution exposure on prediction of placental insufficiency and related outcomes (pre-eclampsia, preterm birth, and IUGR)

CONTACTS AND LOCATIONS:
Overall Officials: Sherin Devaskar, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erickson AC, Arbour L. The shared pathoetiological effects of particulate air pollution and the social environment on fetal-placental development. J Environ Public Health. 2014;2014:901017. doi: 10.1155/2014/901017. Epub 2014 Nov 26. PMID 25574176
- [Background] Liu S, Krewski D, Shi Y, Chen Y, Burnett RT. Association between gaseous ambient air pollutants and adverse pregnancy outcomes in Vancouver, Canada. Environ Health Perspect. 2003 Nov;111(14):1773-8. doi: 10.1289/ehp.6251. PMID 14594630
- [Background] Calkins K, Devaskar SU. Fetal origins of adult disease. Curr Probl Pediatr Adolesc Health Care. 2011 Jul;41(6):158-76. doi: 10.1016/j.cppeds.2011.01.001. PMID 21684471
- [Background] Hricko A. Global trade comes home: community impacts of goods movement. Environ Health Perspect. 2008 Feb;116(2):A78-81. doi: 10.1289/ehp.116-a78. No abstract available. PMID 18288306
- [Background] Su JG, Jerrett M, Beckerman B. A distance-decay variable selection strategy for land use regression modeling of ambient air pollution exposures. Sci Total Environ. 2009 Jun 1;407(12):3890-8. doi: 10.1016/j.scitotenv.2009.01.061. Epub 2009 Mar 21. PMID 19304313
- [Background] Heck JE, Park AS, Qiu J, Cockburn M, Ritz B. Retinoblastoma and ambient exposure to air toxics in the perinatal period. J Expo Sci Environ Epidemiol. 2015 Mar-Apr;25(2):182-6. doi: 10.1038/jes.2013.84. Epub 2013 Nov 27. PMID 24280682
- [Background] Heck JE, Park AS, Qiu J, Cockburn M, Ritz B. An exploratory study of ambient air toxics exposure in pregnancy and the risk of neuroblastoma in offspring. Environ Res. 2013 Nov;127:1-6. doi: 10.1016/j.envres.2013.09.002. Epub 2013 Oct 16. PMID 24139061
- [Background] Heck JE, Park AS, Qiu J, Cockburn M, Ritz B. Risk of leukemia in relation to exposure to ambient air toxics in pregnancy and early childhood. Int J Hyg Environ Health. 2014 Jul;217(6):662-8. doi: 10.1016/j.ijheh.2013.12.003. Epub 2013 Dec 25. PMID 24472648
- [Background] Heck JE, Wu J, Lombardi C, Qiu J, Meyers TJ, Wilhelm M, Cockburn M, Ritz B. Childhood cancer and traffic-related air pollution exposure in pregnancy and early life. Environ Health Perspect. 2013 Nov-Dec;121(11-12):1385-91. doi: 10.1289/ehp.1306761. Epub 2013 Sep 10. PMID 24021746
- [Background] Shrestha A, Ritz B, Wilhelm M, Qiu J, Cockburn M, Heck JE. Prenatal exposure to air toxics and risk of Wilms' tumor in 0- to 5-year-old children. J Occup Environ Med. 2014 Jun;56(6):573-8. doi: 10.1097/JOM.0000000000000167. PMID 24854250
- [Background] Becerra TA, von Ehrenstein OS, Heck JE, Olsen J, Arah OA, Jeste SS, Rodriguez M, Ritz B. Autism spectrum disorders and race, ethnicity, and nativity: a population-based study. Pediatrics. 2014 Jul;134(1):e63-71. doi: 10.1542/peds.2013-3928. PMID 24958588
- [Background] Shah PS, Balkhair T; Knowledge Synthesis Group on Determinants of Preterm/LBW births. Air pollution and birth outcomes: a systematic review. Environ Int. 2011 Feb;37(2):498-516. doi: 10.1016/j.envint.2010.10.009. Epub 2010 Nov 26. PMID 21112090
- [Background] Woodruff TJ, Parker JD, Darrow LA, Slama R, Bell ML, Choi H, Glinianaia S, Hoggatt KJ, Karr CJ, Lobdell DT, Wilhelm M. Methodological issues in studies of air pollution and reproductive health. Environ Res. 2009 Apr;109(3):311-20. doi: 10.1016/j.envres.2008.12.012. Epub 2009 Feb 11. PMID 19215915
- [Background] Aguilera I, Guxens M, Garcia-Esteban R, Corbella T, Nieuwenhuijsen MJ, Foradada CM, Sunyer J. Association between GIS-based exposure to urban air pollution during pregnancy and birth weight in the INMA Sabadell Cohort. Environ Health Perspect. 2009 Aug;117(8):1322-7. doi: 10.1289/ehp.0800256. Epub 2009 Apr 13. PMID 19672415
- [Background] Ballester F, Estarlich M, Iniguez C, Llop S, Ramon R, Esplugues A, Lacasana M, Rebagliato M. Air pollution exposure during pregnancy and reduced birth size: a prospective birth cohort study in Valencia, Spain. Environ Health. 2010 Jan 29;9:6. doi: 10.1186/1476-069X-9-6. PMID 20113501
- [Background] Brauer M, Lencar C, Tamburic L, Koehoorn M, Demers P, Karr C. A cohort study of traffic-related air pollution impacts on birth outcomes. Environ Health Perspect. 2008 May;116(5):680-6. doi: 10.1289/ehp.10952. PMID 18470315
- [Background] Genereux M, Auger N, Goneau M, Daniel M. Neighbourhood socioeconomic status, maternal education and adverse birth outcomes among mothers living near highways. J Epidemiol Community Health. 2008 Aug;62(8):695-700. doi: 10.1136/jech.2007.066167. PMID 18621954
- [Background] Pedersen M, Giorgis-Allemand L, Bernard C, Aguilera I, Andersen AM, Ballester F, Beelen RM, Chatzi L, Cirach M, Danileviciute A, Dedele A, Eijsden Mv, Estarlich M, Fernandez-Somoano A, Fernandez MF, Forastiere F, Gehring U, Grazuleviciene R, Gruzieva O, Heude B, Hoek G, de Hoogh K, van den Hooven EH, Haberg SE, Jaddoe VW, Klumper C, Korek M, Kramer U, Lerchundi A, Lepeule J, Nafstad P, Nystad W, Patelarou E, Porta D, Postma D, Raaschou-Nielsen O, Rudnai P, Sunyer J, Stephanou E, Sorensen M, Thiering E, Tuffnell D, Varro MJ, Vrijkotte TG, Wijga A, Wilhelm M, Wright J, Nieuwenhuijsen MJ, Pershagen G, Brunekreef B, Kogevinas M, Slama R. Ambient air pollution and low birthweight: a European cohort study (ESCAPE). Lancet Respir Med. 2013 Nov;1(9):695-704. doi: 10.1016/S2213-2600(13)70192-9. Epub 2013 Oct 15. PMID 24429273
- [Background] Malmqvist E, Rignell-Hydbom A, Tinnerberg H, Bjork J, Stroh E, Jakobsson K, Rittner R, Rylander L. Maternal exposure to air pollution and birth outcomes. Environ Health Perspect. 2011 Apr;119(4):553-8. doi: 10.1289/ehp.1002564. Epub 2011 Jan 6. PMID 21212043
- [Background] Slama R, Morgenstern V, Cyrys J, Zutavern A, Herbarth O, Wichmann HE, Heinrich J; LISA Study Group. Traffic-related atmospheric pollutants levels during pregnancy and offspring's term birth weight: a study relying on a land-use regression exposure model. Environ Health Perspect. 2007 Sep;115(9):1283-92. doi: 10.1289/ehp.10047. PMID 17805417
- [Background] van den Hooven EH, Jaddoe VW, de Kluizenaar Y, Hofman A, Mackenbach JP, Steegers EA, Miedema HM, Pierik FH. Residential traffic exposure and pregnancy-related outcomes: a prospective birth cohort study. Environ Health. 2009 Dec 22;8:59. doi: 10.1186/1476-069X-8-59. PMID 20028508
- [Background] Wilhelm M, Ritz B. Residential proximity to traffic and adverse birth outcomes in Los Angeles county, California, 1994-1996. Environ Health Perspect. 2003 Feb;111(2):207-16. doi: 10.1289/ehp.5688. PMID 12573907
- [Background] Gehring U, van Eijsden M, Dijkema MB, van der Wal MF, Fischer P, Brunekreef B. Traffic-related air pollution and pregnancy outcomes in the Dutch ABCD birth cohort study. Occup Environ Med. 2011 Jan;68(1):36-43. doi: 10.1136/oem.2009.053132. Epub 2010 Aug 25. PMID 20798012
- [Background] Gehring U, Wijga AH, Fischer P, de Jongste JC, Kerkhof M, Koppelman GH, Smit HA, Brunekreef B. Traffic-related air pollution, preterm birth and term birth weight in the PIAMA birth cohort study. Environ Res. 2011 Jan;111(1):125-35. doi: 10.1016/j.envres.2010.10.004. Epub 2010 Nov 9. PMID 21067713
- [Background] Ritz B, Wilhelm M, Hoggatt KJ, Ghosh JK. Ambient air pollution and preterm birth in the environment and pregnancy outcomes study at the University of California, Los Angeles. Am J Epidemiol. 2007 Nov 1;166(9):1045-52. doi: 10.1093/aje/kwm181. Epub 2007 Aug 4. PMID 17675655
- [Background] Ghosh JK, Wilhelm M, Su J, Goldberg D, Cockburn M, Jerrett M, Ritz B. Assessing the influence of traffic-related air pollution on risk of term low birth weight on the basis of land-use-based regression models and measures of air toxics. Am J Epidemiol. 2012 Jun 15;175(12):1262-74. doi: 10.1093/aje/kwr469. Epub 2012 May 13. PMID 22586068
- [Background] Ritz B. Air pollution and congenital anomalies. Occup Environ Med. 2010 Apr;67(4):221-2. doi: 10.1136/oem.2009.051201. Epub 2009 Nov 2. No abstract available. PMID 19884648
- [Background] Ritz B, Qiu J, Lee PC, Lurmann F, Penfold B, Erin Weiss R, McConnell R, Arora C, Hobel C, Wilhelm M. Prenatal air pollution exposure and ultrasound measures of fetal growth in Los Angeles, California. Environ Res. 2014 Apr;130:7-13. doi: 10.1016/j.envres.2014.01.006. Epub 2014 Feb 8. PMID 24517884
- [Background] Lee PC, Roberts JM, Catov JM, Talbott EO, Ritz B. First trimester exposure to ambient air pollution, pregnancy complications and adverse birth outcomes in Allegheny County, PA. Matern Child Health J. 2013 Apr;17(3):545-55. doi: 10.1007/s10995-012-1028-5. PMID 22544506
- [Background] Ebisu K, Bell ML. Airborne PM2.5 chemical components and low birth weight in the northeastern and mid-Atlantic regions of the United States. Environ Health Perspect. 2012 Dec;120(12):1746-52. doi: 10.1289/ehp.1104763. Epub 2012 Sep 20. PMID 23008268
- [Background] Laurent O, Wu J, Li L, Chung J, Bartell S. Investigating the association between birth weight and complementary air pollution metrics: a cohort study. Environ Health. 2013 Feb 17;12:18. doi: 10.1186/1476-069X-12-18. PMID 23413962
- [Background] Olsson D, Ekstrom M, Forsberg B. Temporal variation in air pollution concentrations and preterm birth-a population based epidemiological study. Int J Environ Res Public Health. 2012 Jan;9(1):272-85. doi: 10.3390/ijerph9010272. Epub 2012 Jan 18. PMID 22470291
- [Background] Proietti E, Roosli M, Frey U, Latzin P. Air pollution during pregnancy and neonatal outcome: a review. J Aerosol Med Pulm Drug Deliv. 2013 Feb;26(1):9-23. doi: 10.1089/jamp.2011.0932. Epub 2012 Aug 2. PMID 22856675
- [Background] Protano C, Scalise T, Orsi GB, Vitali M. A systematic review of benzene exposure during pregnancy and adverse outcomes on intrauterine development and birth: still far from scientific evidence. Ann Ig. 2012 Nov-Dec;24(6):451-63. PMID 23234183
- [Background] Slama R, Thiebaugeorges O, Goua V, Aussel L, Sacco P, Bohet A, Forhan A, Ducot B, Annesi-Maesano I, Heinrich J, Magnin G, Schweitzer M, Kaminski M, Charles MA; EDEN Mother-Child Cohort Study Group. Maternal personal exposure to airborne benzene and intrauterine growth. Environ Health Perspect. 2009 Aug;117(8):1313-21. doi: 10.1289/ehp.0800465. Epub 2009 Apr 1. PMID 19672414
- [Background] Stieb DM, Chen L, Eshoul M, Judek S. Ambient air pollution, birth weight and preterm birth: a systematic review and meta-analysis. Environ Res. 2012 Aug;117:100-11. doi: 10.1016/j.envres.2012.05.007. Epub 2012 Jun 21. PMID 22726801
- [Background] Kliman HJ. Uteroplacental blood flow. The story of decidualization, menstruation, and trophoblast invasion. Am J Pathol. 2000 Dec;157(6):1759-68. doi: 10.1016/S0002-9440(10)64813-4. No abstract available. PMID 11106547
- [Background] Khong SL, Kane SC, Brennecke SP, da Silva Costa F. First-trimester uterine artery Doppler analysis in the prediction of later pregnancy complications. Dis Markers. 2015;2015:679730. doi: 10.1155/2015/679730. Epub 2015 Apr 20. PMID 25972623
- [Background] Moradi M, Salcudean SE, Chang SD, Jones EC, Buchan N, Casey RG, Goldenberg SL, Kozlowski P. Multiparametric MRI maps for detection and grading of dominant prostate tumors. J Magn Reson Imaging. 2012 Jun;35(6):1403-13. doi: 10.1002/jmri.23540. Epub 2012 Jan 20. PMID 22267089
- [Background] Vourganti S, Rastinehad A, Yerram N, Nix J, Volkin D, Hoang A, Turkbey B, Gupta GN, Kruecker J, Linehan WM, Choyke PL, Wood BJ, Pinto PA. Multiparametric magnetic resonance imaging and ultrasound fusion biopsy detect prostate cancer in patients with prior negative transrectal ultrasound biopsies. J Urol. 2012 Dec;188(6):2152-2157. doi: 10.1016/j.juro.2012.08.025. Epub 2012 Oct 18. PMID 23083875
- [Background] Shah V, Turkbey B, Mani H, Pang Y, Pohida T, Merino MJ, Pinto PA, Choyke PL, Bernardo M. Decision support system for localizing prostate cancer based on multiparametric magnetic resonance imaging. Med Phys. 2012 Jul;39(7):4093-103. doi: 10.1118/1.4722753. PMID 22830742
- [Background] Huen I, Morris DM, Wright C, Parker GJ, Sibley CP, Johnstone ED, Naish JH. R1 and R2 * changes in the human placenta in response to maternal oxygen challenge. Magn Reson Med. 2013 Nov;70(5):1427-33. doi: 10.1002/mrm.24581. Epub 2012 Dec 27. PMID 23280967
- [Background] Ozkaynak H, Baxter LK, Dionisio KL, Burke J. Air pollution exposure prediction approaches used in air pollution epidemiology studies. J Expo Sci Environ Epidemiol. 2013 Nov-Dec;23(6):566-72. doi: 10.1038/jes.2013.15. Epub 2013 May 1. PMID 23632992
- [Background] Robson PM, Madhuranthakam AJ, Dai W, Pedrosa I, Rofsky NM, Alsop DC. Strategies for reducing respiratory motion artifacts in renal perfusion imaging with arterial spin labeling. Magn Reson Med. 2009 Jun;61(6):1374-87. doi: 10.1002/mrm.21960. PMID 19319891
- [Background] Wang R, Yu S, Alger JR, Zuo Z, Chen J, Wang R, An J, Wang B, Zhao J, Xue R, Wang DJ. Multi-delay arterial spin labeling perfusion MRI in moyamoya disease--comparison with CT perfusion imaging. Eur Radiol. 2014 May;24(5):1135-44. doi: 10.1007/s00330-014-3098-9. Epub 2014 Feb 21. PMID 24557051
- [Background] Wang DJ, Bi X, Avants BB, Meng T, Zuehlsdorff S, Detre JA. Estimation of perfusion and arterial transit time in myocardium using free-breathing myocardial arterial spin labeling with navigator-echo. Magn Reson Med. 2010 Nov;64(5):1289-95. doi: 10.1002/mrm.22630. PMID 20865753
- [Background] Wang DJ, Alger JR, Qiao JX, Gunther M, Pope WB, Saver JL, Salamon N, Liebeskind DS; UCLA Stroke Investigators. Multi-delay multi-parametric arterial spin-labeled perfusion MRI in acute ischemic stroke - Comparison with dynamic susceptibility contrast enhanced perfusion imaging. Neuroimage Clin. 2013 Jul 6;3:1-7. doi: 10.1016/j.nicl.2013.06.017. eCollection 2013. PMID 24159561
- [Background] Hegde VL, Singh UP, Nagarkatti PS, Nagarkatti M. Critical Role of Mast Cells and Peroxisome Proliferator-Activated Receptor gamma in the Induction of Myeloid-Derived Suppressor Cells by Marijuana Cannabidiol In Vivo. J Immunol. 2015 Jun 1;194(11):5211-22. doi: 10.4049/jimmunol.1401844. Epub 2015 Apr 27. PMID 25917103
- [Background] Wu HH, Gurney PT, Hu BS, Nishimura DG, McConnell MV. Free-breathing multiphase whole-heart coronary MR angiography using image-based navigators and three-dimensional cones imaging. Magn Reson Med. 2013 Apr;69(4):1083-93. doi: 10.1002/mrm.24346. Epub 2012 May 30. PMID 22648856
- [Background] Wu HH, Nishimura DG. 3D magnetization-prepared imaging using a stack-of-rings trajectory. Magn Reson Med. 2010 May;63(5):1210-8. doi: 10.1002/mrm.22288. PMID 20432292
- [Background] Sung K, Hargreaves BA. High-frequency subband compressed sensing MRI using quadruplet sampling. Magn Reson Med. 2013 Nov;70(5):1306-18. doi: 10.1002/mrm.24592. Epub 2012 Dec 27. PMID 23280540
- [Background] Jung H, Sung K, Nayak KS, Kim EY, Ye JC. k-t FOCUSS: a general compressed sensing framework for high resolution dynamic MRI. Magn Reson Med. 2009 Jan;61(1):103-16. doi: 10.1002/mrm.21757. PMID 19097216
- [Background] Sung K, Daniel BL, Hargreaves BA. Location constrained approximate message passing for compressed sensing MRI. Magn Reson Med. 2013 Aug;70(2):370-81. doi: 10.1002/mrm.24468. Epub 2012 Oct 5. PMID 23042658
- [Background] Ritz B, Yu F. The effect of ambient carbon monoxide on low birth weight among children born in southern California between 1989 and 1993. Environ Health Perspect. 1999 Jan;107(1):17-25. doi: 10.1289/ehp.9910717. PMID 9872713
- [Background] Ritz B, Yu F, Fruin S, Chapa G, Shaw GM, Harris JA. Ambient air pollution and risk of birth defects in Southern California. Am J Epidemiol. 2002 Jan 1;155(1):17-25. doi: 10.1093/aje/155.1.17. PMID 11772780
- [Background] Wilhelm M, Ritz B. Local variations in CO and particulate air pollution and adverse birth outcomes in Los Angeles County, California, USA. Environ Health Perspect. 2005 Sep;113(9):1212-21. doi: 10.1289/ehp.7751. PMID 16140630
- [Background] Wu J, Ren C, Delfino RJ, Chung J, Wilhelm M, Ritz B. Association between local traffic-generated air pollution and preeclampsia and preterm delivery in the south coast air basin of California. Environ Health Perspect. 2009 Nov;117(11):1773-9. doi: 10.1289/ehp.0800334. Epub 2009 Jun 23. PMID 20049131
- [Background] Wu J, Wilhelm M, Chung J, Ritz B. Comparing exposure assessment methods for traffic-related air pollution in an adverse pregnancy outcome study. Environ Res. 2011 Jul;111(5):685-92. doi: 10.1016/j.envres.2011.03.008. Epub 2011 Mar 30. PMID 21453913
- [Background] Wilhelm M, Ghosh JK, Su J, Cockburn M, Jerrett M, Ritz B. Traffic-related air toxics and preterm birth: a population-based case-control study in Los Angeles County, California. Environ Health. 2011 Oct 7;10:89. doi: 10.1186/1476-069X-10-89. PMID 21981989
- [Background] Jerrett M, Burnett RT, Beckerman BS, Turner MC, Krewski D, Thurston G, Martin RV, van Donkelaar A, Hughes E, Shi Y, Gapstur SM, Thun MJ, Pope CA 3rd. Spatial analysis of air pollution and mortality in California. Am J Respir Crit Care Med. 2013 Sep 1;188(5):593-9. doi: 10.1164/rccm.201303-0609OC. PMID 23805824
- [Background] Su JG, Jerrett M, Beckerman B, Wilhelm M, Ghosh JK, Ritz B. Predicting traffic-related air pollution in Los Angeles using a distance decay regression selection strategy. Environ Res. 2009 Aug;109(6):657-70. doi: 10.1016/j.envres.2009.06.001. Epub 2009 Jun 21. PMID 19540476
- [Background] Su JG, Jerrett M, Meng YY, Pickett M, Ritz B. Integrating smart-phone based momentary location tracking with fixed site air quality monitoring for personal exposure assessment. Sci Total Environ. 2015 Feb 15;506-507:518-26. doi: 10.1016/j.scitotenv.2014.11.022. Epub 2014 Nov 28. PMID 25437768
- [Background] Schneider R, Haueisen J, Pfeuffer J. Shaped saturation with inherent radiofrequency-power-efficient trajectory design in parallel transmission. Magn Reson Med. 2014 Oct;72(4):1015-27. doi: 10.1002/mrm.25016. Epub 2013 Nov 11. PMID 24408110
- [Background] Avants BB, Epstein CL, Grossman M, Gee JC. Symmetric diffeomorphic image registration with cross-correlation: evaluating automated labeling of elderly and neurodegenerative brain. Med Image Anal. 2008 Feb;12(1):26-41. doi: 10.1016/j.media.2007.06.004. Epub 2007 Jun 23. PMID 17659998
- [Background] Wang J, Alsop DC, Li L, Listerud J, Gonzalez-At JB, Schnall MD, Detre JA. Comparison of quantitative perfusion imaging using arterial spin labeling at 1.5 and 4.0 Tesla. Magn Reson Med. 2002 Aug;48(2):242-54. doi: 10.1002/mrm.10211. PMID 12210932
- [Background] Yan L, Wang S, Zhuo Y, Wolf RL, Stiefel MF, An J, Ye Y, Zhang Q, Melhem ER, Wang DJ. Unenhanced dynamic MR angiography: high spatial and temporal resolution by using true FISP-based spin tagging with alternating radiofrequency. Radiology. 2010 Jul;256(1):270-9. doi: 10.1148/radiol.10091543. PMID 20574100
- [Background] Haas DM, Parker CB, Wing DA, Parry S, Grobman WA, Mercer BM, Simhan HN, Hoffman MK, Silver RM, Wadhwa P, Iams JD, Koch MA, Caritis SN, Wapner RJ, Esplin MS, Elovitz MA, Foroud T, Peaceman AM, Saade GR, Willinger M, Reddy UM; NuMoM2b study. A description of the methods of the Nulliparous Pregnancy Outcomes Study: monitoring mothers-to-be (nuMoM2b). Am J Obstet Gynecol. 2015 Apr;212(4):539.e1-539.e24. doi: 10.1016/j.ajog.2015.01.019. Epub 2015 Jan 31. PMID 25648779
- [Background] Gomez O, Figueras F, Martinez JM, del Rio M, Palacio M, Eixarch E, Puerto B, Coll O, Cararach V, Vanrell JA. Sequential changes in uterine artery blood flow pattern between the first and second trimesters of gestation in relation to pregnancy outcome. Ultrasound Obstet Gynecol. 2006 Nov;28(6):802-8. doi: 10.1002/uog.2814. PMID 17063456
- [Background] Webb E, Bushkin-Bedient S, Cheng A, Kassotis CD, Balise V, Nagel SC. Developmental and reproductive effects of chemicals associated with unconventional oil and natural gas operations. Rev Environ Health. 2014;29(4):307-18. doi: 10.1515/reveh-2014-0057. PMID 25478730
- [Background] Ghosh JK, Heck JE, Cockburn M, Su J, Jerrett M, Ritz B. Prenatal exposure to traffic-related air pollution and risk of early childhood cancers. Am J Epidemiol. 2013 Oct 15;178(8):1233-9. doi: 10.1093/aje/kwt129. Epub 2013 Aug 28. PMID 23989198
- [Background] Beckerman BS, Jerrett M, Serre M, Martin RV, Lee SJ, van Donkelaar A, Ross Z, Su J, Burnett RT. A hybrid approach to estimating national scale spatiotemporal variability of PM2.5 in the contiguous United States. Environ Sci Technol. 2013 Jul 2;47(13):7233-41. doi: 10.1021/es400039u. Epub 2013 Jun 11. PMID 23701364
- [Background] Vanderweele TJ, Arah OA. Bias formulas for sensitivity analysis of unmeasured confounding for general outcomes, treatments, and confounders. Epidemiology. 2011 Jan;22(1):42-52. doi: 10.1097/EDE.0b013e3181f74493. PMID 21052008
- [Background] Arah OA, Chiba Y, Greenland S. Bias formulas for external adjustment and sensitivity analysis of unmeasured confounders. Ann Epidemiol. 2008 Aug;18(8):637-46. doi: 10.1016/j.annepidem.2008.04.003. PMID 18652982
- [Background] Singh P, Le S, Beauchamp RD, Townsend CM Jr, Thompson JC. Inhibition of pentagastrin-stimulated up-regulation of gastrin receptors and growth of mouse colon tumor in vivo by proglumide, a gastrin receptor antagonist. Cancer Res. 1987 Oct 1;47(19):5000-4. PMID 3621187
- [Derived] Lee B, Janzen C, Aliabadi AR, Lei MYY, Wu H, Liu D, Vangala SS, Devaskar SU, Sung K. Early pregnancy imaging predicts ischemic placental disease. Placenta. 2023 Sep 7;140:90-99. doi: 10.1016/j.placenta.2023.07.297. Epub 2023 Jul 31. PMID 37549442